CLINICAL TRIAL: NCT00079573
Title: Benefits & Risks of Popular Weight Loss Diets
Brief Title: Comparison of Popular Weight Loss Diets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Community Foundation of Southeastern Michigan (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT001098-01A1 (NIH)
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Obesity
Keywords: Weight Loss; Obesity; Overweight; Premenopausal women; Diet
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — Diet, High-Protein Low-Carbohydrate

INTERVENTIONS:
Behavioral: Atkins diet (extremely low carbohydrate)
Behavioral: Zone diet (low carbohydrate, high protein)
Behavioral: Ornish diet (very low fat)

SUMMARY:
This study will compare the safety and effectiveness of three popular weight loss plans. These plans will be compared with the USDA Dietary Guidelines.

DETAILED DESCRIPTION:
Obesity is the single most significant, nutrition-related health issue of the new millennium. Several "medical experts" have designed and promoted weight loss diets that dramatically differ from one another and from the USDA Dietary Guidelines. These diets have gained surprisingly widespread and persistent popularity among Americans despite the lack of evidence supporting their claims. This clinical trial will provide preliminary feasibility data for a full-scale study that will examine health outcomes (e.g., benefits, risks, success) of three popular weight loss diets. The study will investigate behavioral and physiological factors that influence adherence and retention to these diet plans.

Overweight women will be randomly assigned to one of four diets for 1 year: Atkins (extremely low carbohydrate), Zone (low carbohydrate, high protein), Ornish (very low fat), or USDA/Food Pyramid (high carbohydrate/moderate-low fat). Behavioral and physiological data will be collected. Participants attend study visits at baseline, 8 weeks, 6 months, and 1 year. At these visits, measurements will include that will include weight and blood pressure measurements and blood tests. Participants will be asked to complete ten questionnaires over the course of the study to assess behavior and appetite. Participants will also undergo a DEXA scan to assess body composition.

ELIGIBILITY:
Inclusion Criteria

* Body mass index (BMI) between 27 and 40 kg/m2
* Weight stable for last 2 months
* Not actively on a weight loss plan
* No plans to move from the area over the next 2 years
* Willing to accept random assignment

Exclusion Criteria

* Pregnant or breastfeeding
* Within 6 months of giving birth or planning to become pregnant in the next 2 years
* Diabetes (type 1 or 2) or history of gestational diabetes
* Renal or liver disease, active neoplasms, or recent myocardial infarction
* Hyper- or hypothyroidism
* Lipid lowering medications or medications known to affect weight/energy expenditure
* Excessive alcohol intake (self-reported, > 3 drinks/day)
* Postmenopausal, including surgical menopause
* Currently under psychiatric care or severely clinically depressed (> 17 on Beck Inventory)

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2002-07; Study Completion 2004-06

PRIMARY OUTCOMES:
Weight; measured at each study visit
Percent body fat; measured at each study visit

SECONDARY OUTCOMES:
Blood lipids (cholesterol, triglycerides); measured at each study visit
Fasting insulin and glucose; measured at each study visit
Behavioral variables; measured at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D. Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Prevention Research Center, Stanford, California, United States

REFERENCES:
- [Derived] Gardner CD, Kiazand A, Alhassan S, Kim S, Stafford RS, Balise RR, Kraemer HC, King AC. Comparison of the Atkins, Zone, Ornish, and LEARN diets for change in weight and related risk factors among overweight premenopausal women: the A TO Z Weight Loss Study: a randomized trial. JAMA. 2007 Mar 7;297(9):969-77. doi: 10.1001/jama.297.9.969. PMID 17341711
- See also: Stanford Center for Research in Disease Prevention — http://prevention.stanford.edu/